CLINICAL TRIAL: NCT03543722
Title: Independence Project: An Intensive Employment Program for Veterans With a Disability Transitioning From the Armed Services
Brief Title: Independence Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Westat (Other)
Collaborators: Tuscaloosa Veterans Affairs Medical Center (U.S. Federal Agency); University of Texas at Austin (Other); Laura and John Arnold Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WPN: 18-148
Record Dates: First submitted 2018-05-02; First posted 2018-06-01 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Employment
Keywords: Veterans; Disability; Employment; Vocational Rehabilitation; Supported Employment

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- National Career Coach Program (Experimental): This program has four main components: a 4-day in-person introductory seminar held in Alpharetta, GA, up to 18 months of job coaching provided by telephone and Skype, a human capital fund to pay for expenses of securing a job (e.g., travel, clothing, computers, professional organization fees), and an opportunity for two years to earn a bonus for employment earnings above a certain level.
  Interventions: Behavioral: National Career Coach Program
- Local Community Resources Program (Active Comparator): Consists of referral to three local face-to-face service providers offering veterans training, financial assistance, and paid work experiences: The Department of Veterans Affairs Compensated Work Therapy Program, the state Vocational Rehabilitation program, and the Department of Labor America's Job Center.
  Interventions: Behavioral: Local Community Resources Program

INTERVENTIONS:
Behavioral: National Career Coach Program — Intensive employment services as described above.
  Arms: National Career Coach Program
Behavioral: Local Community Resources Program — Usual employment services as described above.
  Arms: Local Community Resources Program

SUMMARY:
The Independence Project is a study to evaluate the effectiveness of an intensive employment intervention for young veterans with disabilities recently separated from military service. The study is a randomized controlled trial comparing an intensive employment model (National Career Coach Program) to usual community employment services available to unemployed veterans recently separated from active duty (Local Community Resources Program). The investigators will evaluate if people who receive the National Career Coach Program have better employment outcomes and reduced Veterans Disability Compensation participation than people who receive the Local Community Resources Program.

DETAILED DESCRIPTION:
Tens of thousands of veterans with disabilities transition from military service each year, often destined for lives dependent on disability insurance and disengaged from community life. The personal and societal costs of not helping these veterans re-integrate into civilian life are enormous, including suicides, addiction, family problems, and rapidly increasing costs to the Veterans Disability Compensation Program (VDC).

The current project is an evaluation of the National Career Coach Program to assist veterans as they transition to civilian life. Instead of existing veteran services (including the VDC) that emphasize brokenness and pay veterans small amounts based on what they cannot do, this innovative program emphasizes strengths and abilities by front-loading intensive support, motivation, human-capital investment, and incentives to help veterans become permanently engaged in meaningful work, thereby boosting morale, positive identity, and community integration.

The design of this study is a randomized controlled trial comparing an intensive employment model (National Career Coach Program) to usual community employment services available to unemployed veterans recently separated from active duty (Local Community Resources). The investigators will enroll 250 participants over an 12-month period, randomly assigning them to the two conditions and following them over a three-year period. The primary outcome domains are competitive employment and VDC disability benefits.

ELIGIBILITY:
Inclusion Criteria:

* Former or current US Armed Service members.
* Enlisted rank at time of separation.
* Under 45 years old.
* Completed at least six months of active duty.
* Received or will receive honorable or general discharge.
* At time of enrollment, their Expiration of Term of Service is within six months prior to separation or within 12 months post-separation.
* Completed an application for a Veterans Disability Compensation (VDC) rating and waiting determination, or, if the VDC rating has been determined, awarded a disability rating between 30% to 90%.
* If currently on active duty, no intention to reenlist or to accept an existing offer for a permanent job upon separation; if already separated from active duty, currently unemployed (or employed in temporary job).
* Expressed desire to work in a competitive job within 3 months of separation (if on active duty) or within 3 months (if separated from active duty).
* Willing to participate in either of the two employment approaches including attendance at a scheduled introductory class.
* Consent to research procedures.

Exclusion Criteria:

• None

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Earnings | 36 months
  Amount earned from competitive employment as reported by IRS administrative earnings data
Veterans Disability Compensation rating and benefits | 36 months
  Department of Veterans Affairs Schedule for Rating Disabilities, which assigns a percentage from 0% to 100%, the higher the value the more significant the disability

CONTACTS AND LOCATIONS:
Overall Officials: Gary R Bond, PhD, Principal Investigator — Westat; Robert E Drake, PhD, Principal Investigator — Westat
Locations (1):
- Westat, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No